CLINICAL TRIAL: NCT04428047
Title: A Phase II Trial Assessing Bintrafusp Alfa, a Bifunctional Fusion Protein Targeting TGF-β and PD-L1, in a Pre-operative Setting for Resectable and Untreated Head and Neck Squamous Cell Carcinoma
Brief Title: Evaluation of Bintrafusp Alfa in Operable and Untreated Head and Neck Squamous Cell Carcinoma
Acronym: ICING
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision following information on cases of hyperprogression and early toxicities with bintrafusp alfa in other studies
Sponsor: UNICANCER (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC-HNG/1909; 2019-004052-11 (EudraCT Number)
Record Dates: First submitted 2020-06-02; First posted 2020-06-11 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
Keywords: PDL1 blockade; TGFb trap; PathR; window-of-opportunity preoperative trial
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — bintrafusp alfa protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- bintrafusp alfa (Experimental): bintrafusp alfa will be administered by intravenous infusion over 60 minutes at a dose of 1200 mg on Day1 and Day15
  Interventions: Drug: bintrafusp alfa

INTERVENTIONS:
Drug: bintrafusp alfa — bintrafusp alfa will be administered by intravenous infusion over 60 minutes at a dose of 1200 mg on Day1 and Day15
  Other Names: M7824

SUMMARY:
This study is a prospective open label, multicenter, phase II, window-of-opportunity preoperative, single-agent trial.

This study aims to evaluate the efficacy, the safety and tolerability profile of bintrafusp alfa in patients with histologically or cytologically confirmed squamous cell carcinoma of the oral cavity, oropharynx, larynx or hypopharynx, previously untreated, with indication of primary surgery. Patients with a diagnosis of head and neck squamous cell carcinoma (HNSCC) from unknown primary will not be enrolled.

DETAILED DESCRIPTION:
The study plans to enrol up to 59 patients in total. Eligible patients who have provided their written informed consent for study participation will be assigned to one the 2 cohorts described below:

Cohort A (43 patients): Non-oropharyngeal HNSCC, or Oropharyngeal squamous cell carcinoma (SCC) that are human papillomavirus (HPV) negative, or Oropharyngeal SCC that are HPV positive and smoker ≥20 pack year (PY).

A Minimax two-stage Simon design will be used with an unacceptable rate of pathological response of 30% or less and a hypothesized actual pathological response rate of 50% or more.

In the first stage, 28 patients will be accrued. If the observed number of patients with a pathological response is 7 or less, then the study for the cohort A will conclude to inefficacy and patient recruitment in this cohort will be stopped.

Cohort B (16 patients): Oropharyngeal SCC that are HPV positive and non-smoker or smoker <20 PY (former or active).

The design for this cohort will be a single-stage design.

All trial-related interventions will be strictly similar for these 2 cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Patients must have signed a written informed consent form prior to any trial specific procedures
3. Histologically or cytologically confirmed HNSCC of the oral cavity, oropharynx, larynx or hypopharynx, previously untreated, with indication of primary surgery. Patients with a diagnosis of HNSCC of occult primary could not be enrolled.

   In order to avoid repeated biopsies procedures under general anesthesia, patients with clinically highly suspected squamous cell carcinoma could be registered before the histological or cytological proof. In these cases, the diagnosis will be confirmed rapidly after the endoscopy, either by using frozen sections or by reporting the results obtained on formalin-fixed paraffin-embedded (FFPE) within no more than 5 working days.
4. Absence of distant metastases determined by CT-scan or PET-CT that must be performed within 35 days prior to endoscopy.
5. According to the 7th edition American Joint Committee on Cancer (AJCC) eligible stages are as follow:

   T2N1, T2N2, T2N3 T3 or T4 (any N)
6. Baseline radiology studies evaluating primary tumor (MRI or CT-scan) must be performed within 28 days prior to endoscopy.
7. Patients must have at least 1 lesion superior to 2 cm in larger axis
8. Eastern Cooperative Oncology Group (ECOG) performance status ≤1
9. Adequate organ and marrow function as defined by the following laboratory results obtained within 28 days prior to the baseline endoscopy:

   1. Hemoglobin (Hb) ≥9,0 g/dL;
   2. Absolute neutrophil count (ANC) ≥1,500/mm³;
   3. Platelet count ≥100,000/mm³;
   4. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤1.5 × institutional upper limit of normal (ULN);
   5. Total bilirubin ≤1.5 × ULN;
   6. Creatinine clearance >30 mL/min as determined by the Cockcroft-Gault equation (Cockcroft and Gault, 1976)
10. Negative serology for hepatitis B and C
11. Patients must be willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures
12. Willing and able to provide tumor specimen and blood samples for translational research.
13. Women of childbearing potential must have a negative serum β-human chorionic gonadotropin (β-HCG) pregnancy test within 7 days prior to the administration of the first study treatment and/or urine pregnancy 48 hours prior to the administration of the first study treatment.
14. Both sexually active women of childbearing potential and males (and their female partners) patients must agree to use two methods of effective contraception, one of them being a barrier method, or to abstain from sexual activity during the study and for at least 2 months after last dose of study drugs.
15. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
16. Patients must be affiliated to the social security system or equivalent

Exclusion Criteria:

1. Primary site of head and neck carcinoma in nasopharynx, sinuses, or skin
2. Patients receiving other anti-cancer medication such as, chemotherapy, immunotherapy, biologic therapy, targeted therapy, monoclonal antibodies, hormonal therapy (other than leuprolide or other gonadotropin releasing hormone (GnRH) agonists) or other investigational agent within 6 months prior to the first dose of study drug and while on study treatment.
3. Patients receiving other anti-cancer non-drug therapies: radiation, or tumor embolization within 6 months prior to the first dose of study drug and while on study treatment.
4. Previous or concurrent cancer within 2 years prior to study inclusion including symptomatic, untreated, or actively progressing central nervous system (CNS) metastases, with the exception of the following cancer types: in situ carcinomas of any location; skin basal cell carcinoma stage T1N0M0 or T2N0M0
5. Any previous treatment with a PD-1, PD-L1 agent
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, active peptic ulcer disease or gastritis, active bleeding diatheses.
7. Current or prior use of immunosuppressive medication within 28 days before the first dose of bintrafusp alfa, with the exceptions of intranasal, intraocular and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone or an equivalent corticosteroid.
8. Receipt of live attenuated vaccination within 28 days prior to the first administration of bintrafusp alfa.
9. History of (non-infectious) pneumonitis that required steroids within 28 days prior to the first administration of bintrafusp alfa or current pneumonitis.
10. Major surgery within 28 days prior to the first administration of bintrafusp alfa and not recovered adequately from the toxicities and/or complications.
11. Serious, non-healing or dehiscing, wound, active ulcer, or ongoing bone fracture.
12. Active or prior documented autoimmune disease within the past 2 years. Note: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) can be enrolled
13. Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
14. History of primary immunodeficiency
15. History of allogenic organ transplant that requires the use of immunosuppressive drugs
16. Pregnant or breast-feeding women
17. Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
18. Known positive HIV status
19. Participation in another clinical study with an investigational product during the last 28 days.
20. Known hypersensitivity to the study drug, study drug classes, or study drug excipients.
21. Patients under guardianship or deprived of his liberty by a judicial or administrative decision or any condition (e.g., psychiatric illness/social/familial/geographical condition) that would limit compliance with study requirement or compromise the ability of the patients to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2021-09-04 (Actual); Study Completion 2022-01-07 (Actual)

PRIMARY OUTCOMES:
Pathological response (PathR) | From inclusion to 1 month after surgery
  Pathological tumor response will be evaluated as the percentage of the tumor area showing evidence of anti-tumor activity, such as tumor cell necrosis and/or giant cell/histolytic reaction to keratinous debris

SECONDARY OUTCOMES:
Pathological response using a threshold of 50% (PathR50), 70% (PathR70) and 90% (PathR90) | From inclusion to 1 month after surgery
  Will be considered as responders, the patients presenting 50% or more, 70% or more, and 90% or more, respectively, of tumor cell death.
Response rate, using primary endpoint criteria, by PD-L1 status | 3 years
  The response rate using primary endpoint criteria, by PD-L1 status using Combined Positive Score (CPS) thresholds of 1 and 20. CPS is the number of PD-L1 staining cells (tumor cells and immune cells) divided by the total number of viable tumor cells, multiplied by 100.
Response rate, using primary endpoint criteria, by HPV status in cohort A | 2 years
  The response rate, using primary endpoint criteria, by HPV status determined by p16 staining in cohort A. Two categories will be defined: HPV- and HPV+ (smokers ≥20 PY). HPV+ non-smoker or smoker <20 PY will be included in cohort B.
Clinical response | From inclusion to post-treatment imaging visit, an average of 21 days
  Efficacy of bintrafusp alfa by clinical response will be evaluated by measuring changes in tumor size in response to treatment; measured by Magnetic resonance Imaging (MRI) or positron emission tomography (PET) scan and assessed by RECIST v1.1
Disease-free survival (DFS) | 12, 18, 24, and 36 months after surgery
  DFS defined as the delay between the date of the surgery and the occurrence of a loco-regional recurrence and/or a distant metastasis due to the cancer or death whatever the cause for which the patient was included, whichever comes first.
Overall survival (OS) | 12, 18, 24, and 36 months after surgery
  OS defined as the delay between the date of the surgery and the occurrence of death, whatever the cause.
Loco-regional disease-free survival (LR-DFS) | 12, 18, 24, and 36 months after surgery
  LR-DFS defined as the delay between the date of the surgery and the first occurrence of a loco-regional recurrence due to the cancer or death whatever the cause for which the patient was included.
Distant disease-free survival (D-DFS) | 12, 18, 24, and 36 months after surgery
  D-DFS defined as the delay between the date of the surgery and the first occurrence of a distant metastasis due to the cancer or death whatever the cause for which the patient was included.
Treatment-Emergent Adverse Events (Safety and Tolerability) profile of bintrafusp alfa | From inclusion to 12 weeks after the last administration of the investigational product
  The National Cancer Institute-Common Terminology Criteria for Adverse Events version 5 (NCI-CTCAE v5) is widely accepted in the community of oncology research as the leading rating scale for adverse events. This scale will assess the severity of sensory neuropathic disorders, this derivative into 5 grades determined by the investigator.
Evaluation of the impact of inking the tumor margins during baseline endoscopy to avoid surgical plan changes putatively induced by tumor shrinking under therapy | From inclusion to surgery, an average of 21 days
  Just before the beginning of the surgery, surgeons will answer a question (4-level: Yes, No, Not evaluable, Unknown) to indicate if their surgical plan would have been different in the absence of ink labelling.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Hoffmann, MD, PhD, Principal Investigator — Institut Curie; Christophe Letrouneau, MD, PhD, Principal Investigator — Institut Curie
Locations (8):
- France (8):
  - CHU de Bordeaux, Bordeaux
  - Centre Antoine Lacassagne, Cagnes-sur-Mer
  - Centre Léon Bérard, Lyon
  - CHU La Timone, Marseille
  - Institut Curie, Paris
  - Institut Claudius Régaud, Toulouse
  - Institut de cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Gustave Roussy Cancer Campus, Villejuif

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients.

REFERENCES:
- [Derived] Saint A, Van Obberghen-Schilling E. The role of the tumor matrix environment in progression of head and neck cancer. Curr Opin Oncol. 2021 May 1;33(3):168-174. doi: 10.1097/CCO.0000000000000730. PMID 33720067